CLINICAL TRIAL: NCT06928038
Title: The Effect of Maternal Position on Labour Progression in Deliveries With the Foetus in the Occiput Posterior Position
Brief Title: Maternal Position's Effect on Labor Progression in Occiput Posterior Deliveries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Nezihe KIZILKAYA BEJI, Professor, Biruni University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10840098-241
Record Dates: First submitted 2025-03-28; First posted 2025-04-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Labor; Prolonged, Second Stage; Delivery Problem
Keywords: Foetal malposition; Occiput posterior stance; Delivery positions
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Intervention Model Description: The study included 148 gravidas admitted to a private Istanbul hospital, who consented to participate. They were divided into intervention and control groups (n=72). The intervention group assumed a side-lying position on the occiput side for 20 minutes, a prostrate position for 15 minutes, then leaned towards the bed's head for 10 minutes (rest), followed by another 20-minute side-lying position. The control group received routine delivery care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The positioned group assumed a side-lying position on the occiput side for 20 minutes, a prostrate position for 15 minutes, then leaned towards the bed's head for 10 minutes (rest), followed by another 20-minute side-lying position.
  Interventions: Behavioral: Positioned group
- Control group (No Intervention): The control group was followed up in the routine delivery room, and no positioning was done.

INTERVENTIONS:
Behavioral: Positioned group — applied a side-lying position (20 minutes) on the occiput side and a prostrate position (15 minutes).
  Arms: Intervention group

SUMMARY:
This is a randomized controlled experimental study to determine the effect of maternal position on the progression of labour in deliveries in which the foetus is in the occiput posterior position.

The study included 148 gravidas admitted to a private Istanbul hospital, who consented to participate. They were divided into intervention and control groups (n=72). The intervention group assumed a side-lying position on the occiput side for 20 minutes, a prostrate position for 15 minutes, then leaned towards the bed's head for 10 minutes (rest), followed by another 20-minute side-lying position. The control group received routine delivery care.

DETAILED DESCRIPTION:
This is a randomized controlled experimental study. The research was carried out in a private hospital in Istanbul. The population of the study covered gravidas who were admitted to the hospital for delivery with the foetus in the occiput posterior position in labour. The sample of the study included 148 volunteering gravidas, who were divided into intervention and control groups.

Research Hypotheses:

H1: In deliveries where the foetus is in the occiput posterior position, the positions given to the mother help the foetus to rotate to the occiput anterior position.

H2: Positions given to the mother in the occiput posterior position do not affect the Apgar score.

H3: In deliveries where the foetus is in the occiput posterior position, the positions given to the mother reduce the rate of interventional delivery.

Implementation :

After the occiput posterior position was established by ultrasonography, the gravidas included in the study were randomized into 2 groups as intervention and control groups. The intervention group was given the following positions during labour:

1. The gravida is given a side-lying position on the side of the occiput for 20 minutes. She is laid with the lower leg bent and the upper leg extended.
2. Then the prostrate position is given for 15 minutes (This position is where the pregnant women kneels while lowering her forehead to touch the bed or floor).
3. After this position, they are allowed to rest for 10 minutes by leaning towards the head of the bed.
4. Then, they are given a side-lying position again on the side of the occiput for 20 minutes.

After 1 hour, the gravida was placed in a side lying position on the side of the occiput. Digital vaginal examination was repeated at 2 hour intervals. If the foetus has rotated to the occiput anterior position, the women was released (could walk, stand, allowed to do as she pleased). If the occiput posterior continued but the descent of the head was progressing, she was tilted to the side of the occiput on the delivery table after the dilatation is completed and instructed to push (keeping the upper leg up). At the time of coronation, she was laid on her back and delivered. If there was no head descent or rotation according to the digital vaginal examination finding, time was allowed for dilatation to reach 7-8 cm in the primiparae. Caeserean section (C/S) was scheduled if there was no change. If the posh was not open in multiparous patients and the head was at -3 -2, amniotomy was performed and time was allowed until dilatation was complete. However, C/S was planned if digital vaginal examination performed with an interval of 2 hours did not indicate progress.

The control group was followed up in the routine delivery room, and no positioning was done.

ELIGIBILITY:
Inclusion Criteria:

* Gravidas aged 18 years or older
* Between 36 and 42 weeks of gestation
* Willing to participate in the study
* Expected to deliver vaginally
* Not classified as high-risk
* No obstetric or medical complications during labor
* Single, healthy fetus in one of the following positions: occiput posterior, left occiput posterior, right occiput posterior, left occiput transverse, or right occiput transverse (confirmed via ultrasonography)
* Cervical dilation of at least 2-3 cm
* Estimated fetal weight between 2500 g and 3999 g
* No major congenital anomalies

Exclusion criteria:

Inability to understand Turkish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
birth type of the baby | from labor to the end of the delivery
  cesarean section, spontaneously deliver
Head position | From labor to the expulsion stage
  right - left occiput posterior; right - left occiput transverse; right - left occiput anterior

SECONDARY OUTCOMES:
duration of expulsion phase | duration of expulsion phase
  The time from completion of dilatation to birth of the baby